CLINICAL TRIAL: NCT05441644
Title: Comparative Study of Bispectral Index (BIS) Values Obtained From Standard Frontal Position and Alternative Infra-orbital Position During Total Intravenous Anaesthesia (TIVA).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohamad Hasyizan Hassan, Senior Lecturer and Neuroanaesthesiologist, Universiti Sains Malaysia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: USM/JEPeM/20060307
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Intraoperative Awareness
MeSH Terms: conditions — Intraoperative Awareness | interventions — Consciousness Monitors

STUDY DESIGN:
Intervention Model Description: two way mixed effect model; aggreement study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- frontal BIS (Placebo Comparator): frontal BIS is a standard position
  Interventions: Device: Bispectral index
- infraorbital BIS (Active Comparator): Infraorbital BIS is a comparator to find agreement with standard location
  Interventions: Device: Bispectral index

INTERVENTIONS:
Device: Bispectral index — A new placemewnt to monitor intraoperative BIS

SUMMARY:
A study to find agreement of the infraorbtal BIS placement as compared to standard frotal placement

DETAILED DESCRIPTION:
2.1 Study Design This was a prospective, cross-sectional study conducted in single centre, University Hospital. The study protocol was reviewed and granted approval for implementation by the institution Human Research and Ethics Committee (study protocol code: USM/JEPeM/20060307).

2.2 Study Population We recruited 71 patients who were eligible to be enrolled in this study from November 2020 to October 2021. The inclusion criteria were consented adults between the age of 18 and 60 years old, BMI > 18 and <30 kg/m2 and ASA physical status I or II underwent general elective surgery under general anaesthesia. We excluded patients who were going for neurosurgery, maxillofacial or facial surgical procedures because the operation site may interfere with the BIS sensors placement. Patients with a history of disabling central nervous or cerebrovascular disease, those on psychiatric medication or central nervous system active drugs, and those who had undergone neurosurgical procedure were also excluded. The patient who had interruption of BIS monitoring of any BIS sensor location at any time frame will be withdrawn from the study.

The baseline demographic data of patients were extracted from their medical chart. Demographic data include their age, gender, BMI, ASA physical status and type of surgery.

2.3 Study Method Before induction of anaesthesia, we applied two BIS sensors on each patient at different location (frontal & infra-orbital) and connected two different BIS monitor. Frontal sensors were applied with circle 1 at the centre of forehead, circle 2 2.8cm lateral to circle 1, circle 3 on the corner of the eye and circle 4 in between circle 2 and circle 3 (Picture 1(A)). Infra-orbital sensors were applied with circle 1 across the nose bridge, circle 2 adjacent to circle 1, circle 3 medial from the frontally placed third electrode and circle 4 in between circle 2 and 3 (Picture 1 (B)). Anaesthesia was induced with TCI remifentanil at initial target concentration at 2ng/ml up to 4ng/ml followed with TCI propofol at initial target concentration at 4mcg/ml then titrated upwards to loss of consciousness and intravenous (IV) rocuronium 1.0 mg/kg for muscle relaxant and endotracheal intubation. Anaesthesia was maintained with propofol infusion at target plasma concentration of 3-6mcg/ml and remifentanil 1-8ng/ml; Intra-operative analgesia included IV paracetamol 1g, IV parecoxib 40mg and IV morphine 0.05-0.1mg/kg. At the end of surgery, patients were reversed with IV neostigmine 0.05 mg/kg and atropine 0.02mg/kg. BIS values from each BIS monitor during awake, at loss of consciousness (LOC), after intubation, after the start of surgical incision, every 30 minutes during the intraoperative period (maintenance), after cessation of TCI propofol at which the plasma concentration of propofol is 1.5mcg/ml (emergence) and at extubation were recorded. The frontal BIS was used to guide the depth of anaesthesia, with deep (BIS < 45), moderate (BIS 45 to 60) and mild hypnosis (BIS >60).

2.4 Sample Size In order to determine the Kappa agreement for Pearson's correlation between BIS values obtained from frontal versus the infra-orbital sensor position, using t-test, the sample size would be determined with parameter of effect 0.3, an alpha of 0.05 and a power of 80%. The sample size required was 64 patients and with the estimation of 10% drop-out rate, the total number would be 71 patients.

In order to determine the relationship between BIS values obtained from frontal versus the infra-orbital sensor position, using linear regression, the sample size would be determined with parameter of effect size 0.15, an alpha of 0.05 and a power of 80%. The sample size required was 55 patients.

To satisfy both outcomes, the final sample size for this study would be 71 patients.

2.5 Statistical Analysis Data were recorded and analyzed using SPSS for Window version 22.0. Descriptive statistics were used to summarize the socio-demographic characteristics of subjects. Numerical data were presented as mean (SD) or median (IQR) based on their normality distribution. Categorical data were presented as number and percentage. Correlation of the numerical data obtained from the two different groups were analyzed using Pearson's correlation and scatter plot analysis. Relationship between data obtained from the two groups was determined using simple linear regression.

ELIGIBILITY:
The inclusion criteria were consented adults between the age of 18 and 60 years old, BMI > 18 and <30 kg/m2 and ASA physical status I or II underwent general elective surgery under general anaesthesia. We excluded patients who were going for neurosurgery, maxillofacial or facial surgical procedures because the operation site may interfere with the BIS sensors placement. Patients with a history of disabling central nervous or cerebrovascular disease, those on psychiatric medication or central nervous system active drugs, and those who had undergone neurosurgical procedure were also excluded. The patient who had interruption of BIS monitoring of any BIS sensor location at any time frame will be withdrawn from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
agreement between frontal BIS vs infraorbital BIS | intraoperative
  measurements of BIS values on both placement

SECONDARY OUTCOMES:
correlation between frontal BIS vs infraorbital BIS | intraoperative
  to find correlation between both measurement

CONTACTS AND LOCATIONS:
Locations (1):
- School Of Medical Sciences, Health Campus, Universioti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
there will be upcoming research related to current research